CLINICAL TRIAL: NCT00988611
Title: Novel Predictors of ART Outcomes
Brief Title: Assisted Reproductive Technology (ART) Predictors Study
Acronym: ART
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: ART Predictors Study
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Reproductive Aging
Keywords: Reproductive aging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Telomere length assay
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Women undergoing IVF/ART cycles at OU Physicians Reproductive Health Clinic in Oklahoma City, Oklahoma — Women undergoing an IVF/ART treatment cycle at OU Physicians Reproductive Health Clinic in Oklahoma City, Oklahoma, age range 18-44 years old

SUMMARY:
The goals of this research proposal are to further our understanding of the reproductive aging process in women and to improve our ability to clinically assess and model reproductive aging. Reproductive aging is a continuous process that begins many years prior to menopause. Women in their late 30s and early 40s usually maintain normal menstrual function and ovulatory status, yet fertility in these women is considerably compromised compared to younger women. The primary mechanism of reproductive aging is through the process of ovarian primordial follicle (egg) depletion, a process that exhibits considerable variation between women. As a result, the age at which an individual begins to experience infertility and menstrual cycle changes secondary to follicle depletion also varies significantly and is difficult to predict. The clinical assessment of the number of primordial follicles remaining in the ovary has traditionally relied upon the measurement of ovarian or pituitary hormones such as FSH, estradiol, and inhibin B. Unfortunately, these measures are all indirect and poorly sensitive in the assessment of ovarian reserve. More recently, serum levels of anti-Müllerian hormone (AMH) and the ovarian antral follicle count have been utilized as clinical measures of ovarian reserve. Both have been correlated with chronological age and have some predictive power in determining stimulation quantity (the number of oocytes obtained at the time of egg-recovery) in in-vitro fertilization (IVF) treatment cycles. Reproductive aging in women; however, is more than just the depletion of oocytes from a woman's ovaries, but also involves a decline in oocyte quality. The predictive value of these clinical markers of ovarian reserve with regards to oocyte quality is unknown. Additionally, new tools developed to assess biological aging in other organ systems such as white blood cell telomere length and the measurement of advanced glycation end products (AGEs) through skin autofluorescence have not been evaluated with respect to the reproductive aging process. This proposal seeks to develop better models of normal female reproductive aging by identifying novel markers of ovarian reserve and determining their relationship with both oocyte quantity and quality obtained during IVF treatment cycles.

DETAILED DESCRIPTION:
To test our hypotheses, we will enroll 120 healthy women undergoing ART cycles at OU Physicians Reproductive Health.

Patients undergoing an ART treatment cycle at the OU Physicians Reproductive Health clinic will be approached regarding enrollment.

* informed consent
* collection of baseline demographic data (height, weight, ethnicity, age)
* cycle-day 3 measurements of FSH, estradiol, inhibin B, AMH, white-blood cells for telomere length assay, and measurement of hemoglobin A1C to control for blood glucose levels
* AFC as determined by transvaginal ultrasound exam
* skin autofluorescence measurement
* subjects then undergo IVF as directed by their physician
* outcome measures include number of oocytes recovered, peak estradiol, quantity of gonadotropins utilized during the course of treatment, and assessment of oocyte quality by morphology assessment with light microscopy.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing an ART treatment cycle
* Age range 18-44 years old

  * NOTE: Must be willing to travel to Oklahoma City to participate. Need to have the transvaginal ultrasound and skin autofluorescence measurement at the OU Physicians Reproductive Health Clinic in Oklahoma City, Oklahoma
  * NOTE: Study will not pay for ART/IVF treatment.

Exclusion Criteria:

* Gynecological malignancy
* chemotherapy or radiation therapy treatment
* Autoimmune disease
* Prior ovarian surgery
* Ovarian pathology

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing an ART treatment cycle at the OU Physicians Reproductive Health clinic in Oklahoma City, Oklahoma will be approached regarding enrollment.
  NOTE: Must be willing to travel to Oklahoma City to participate. Need to have the transvaginal ultrasound and skin autofluorescence measurement at the OU Physicians Reproductive Health Clinic in Oklahoma City, Oklahoma
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Determine whether newly described measures of biological age and oxidative stress (white-blood cell telomere length and AGEs measured by skin autofluorescence) are correlated with stimulation quantity (number of oocytes retrieved) in IVF cycles. | 2 years

SECONDARY OUTCOMES:
Determine whether white blood cell telomere length and AGEs measured by skin autofluorescence are correlated with oocyte quality in IVF cycles after adjustment for chronological age. | 2 years
Determine whether established clinical markers of quantitative ovarian reserve (AMH, AFC, FSH, and inhibin B) are correlated with oocyte quality in IVF cycles after adjustment for chronological age. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Karl R Hansen, MD, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States